CLINICAL TRIAL: NCT04514016
Title: Cross Sectional Survey Of Severe Acute Respiratory Syndrome (SARS) Coronavirus 2 (COV-2) Infection And Seroprevalence In A Cohort Of HIV-Infected Children, Youth, And Adolescents
Brief Title: Cross Sectional CFAR HIV/COVID-19 Study
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: Miami Center for AIDS Research (CFAR) (Unknown)
Responsible Party: Principal Investigator, Charles Mitchell, Professor, University of Miami
Other Study IDs: 20200802
Record Dates: First submitted 2020-08-13; First posted 2020-08-14 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: SARS-CoV Infection; Covid19
Keywords: HIV
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, Nasopharyngeal swab samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV positive participants with positive COVID-19 results: Participants in this group will have a RT-PCR and Coronavirus Disease (COVID) -19 specific antibody testing at baseline, 1 month and 3 month visits.
- HIV positive participants with negative COVID-19 results: Participants in this group will have a RT-PCR and COVID-19 specific antibody testing at baseline only.

SUMMARY:
The main purpose of this research study is to learn the rate of SARS COV-2 on HIV infected children, adolescents, and youth receiving their primary HIV care at the University of Miami Miller School of Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Being a patient to the Pediatric or Adolescent clinic located at Batchelor Children Research Institute (BCRI)
* Being diagnosed with HIV infection by the time of enrollment
* At enrollment, 3 to < 26 years

Exclusion Criteria:

* Patient will be excluded from the study if any of the following are identified:
* Patients under legal age and in the State's custody
* Participant or legal guardian unable to sign Informed Consent forms
* Participant unable to complete study visits

Ages: 3 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: HIV-positive pediatric, adolescent or young adult being treated at Batchelor Children Research Institute (BCRI) at the University of Miami.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Number of participants who tested positive with SARS COV-2 Infection | month 3
  SARS COV-2 Infection will be analyzed from nasopharyngeal swab samples via RT-PCR assay
Number of participants who tested positive with SARS COV-2 antibody | month 3
  SARS COV-2 antibody will be analyzed from blood samples via serological assay

CONTACTS AND LOCATIONS:
Overall Officials: Charles Mitchell, MD, Principal Investigator — University of Miami
Locations (1):
- Batchelor's Children's Research Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No